CLINICAL TRIAL: NCT00686218
Title: A Phase I Dose Escalation Study of LBH589 in Combination With Imatinib Mesylate for Patients With Chronic Myeloid Leukemia in Cytogenetic Remission With Residual Disease Detectable by Q-PCR
Brief Title: Panobinostat (LBH589) and Imatinib Mesylate in Treating Patients With Previously Treated Chronic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07203; P30CA033572 (NIH); NOVARTIS-CSTI571AUS275T; CDR0000596065 (Registry Identifier: PDQ); NCI-2010-00528 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-05-28; First posted 2008-05-29 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase | interventions — Imatinib Mesylate; Panobinostat; Polymerase Chain Reaction; Blotting, Western; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (panobinostat, imatinib mesylate) (Experimental): Patients receive oral panobinostat once daily on days 1, 3 and 5; 8, 10, and 12; 15, 17, and 19; and 22, 24, and 26. Patients also receive oral imatinib mesylate once daily on days 1-28. Treatment repeats every 21 or 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Drug: panobinostat; Genetic: polymerase chain reaction; Genetic: protein expression analysis; Genetic: western blotting; Other: flow cytometry; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Drug: panobinostat — Given orally
  Other Names: Faridak; HDAC inhibitor LBH589; histone deacetylase inhibitor LBH589; LBH589
Genetic: polymerase chain reaction — Testing
Genetic: protein expression analysis — Testing
Genetic: western blotting — Testing
Other: flow cytometry — Testing
Other: laboratory biomarker analysis — Testing
Other: pharmacological study — Testing

SUMMARY:
RATIONALE: Panobinostat and imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of panobinostat when given together with imatinib in treating patients with previously treated chronic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety and tolerability of LBH589 given in combination with imatinib mesylate in CML patients who are in Major Cytogenetic Remission (MCR) with residual BCR-ABL positive cells after at least 1 year of daily imatinib mesylate treatment.
* To determine the maximum tolerated dose (MTD) and dose-limiting toxicity of LBH589 given in combination with imatinib mesylate in CML patients.

Secondary

* To study the effect of LBH589 given in combination with imatinib mesylate on cytogenetic response status and BCR-ABL levels in CML patients in major cytogenetic remission on imatinib mesylate treatment.

Tertiary

* To study the effect of LBH589 given in combination with imatinib mesylate on residual BCR-ABL positive primitive progenitors in CML patients in major cytogenetic remission on imatinib mesylate treatment.

OUTLINE: This is dose-escalation study of panobinostat.

Patients receive oral panobinostat once daily on days 1, 3 and 5; 8, 10, and 12; 15, 17, and 19; and 22, 24, and 26. Patients also receive oral imatinib mesylate once daily on days 1-28. Treatment repeats every 21 or 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 month and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* CML CP patients who have been treated with and tolerated Imatinib for 1 year or more, have achieved at least major cytogenetic response and continue to be BCR-ABL positive (Patients should be receiving Imatinib at a dose of 400 daily at the time of entry into the study)
* ANC and PLT need to be in the normal range
* Serum albumin >= 3g/dL
* AST/SGOT and ALT/SGPT =< 2.5 x upper limit of normal (ULN)
* Serum bilirubin =< 1.5 x ULN
* Serum creatinine =< 1.5 x ULN or 24-hour creatinine clearance >= 50 ml/min
* Serum potassium >= lower limit of normal (LLN)
* Serum phosphorus >= LLN
* Serum total calcium (corrected for serum albumin) or serum ionized calcium >= LLN
* Serum magnesium >= LLN
* ECOG performance status of =< 2

Exclusion Criteria:

* Prior treatment with an HDAC inhibitor
* Patient who have been treated with Imatinib < 1 year or patients are currently being treated with Imatinib at a dose > 400 mg daily
* Impaired cardiac function including any one of the following: Screening ECG with a QTc > 450 msec; Patients with congenital long QT syndrome; History or presence of sustained ventricular tachycardia; Any history of ventricular fibrillation or torsades de pointes; Bradycardia defined as heart rate < 50 beats per minute (patients with a pacemaker and heart rate >= 50 beats per minute are eligible); Patients with a myocardial infarction or unstable angina within 6 months of study entry; Congestive heart failure (NY Heart Association class III or IV); Right bundle branch block and left anterior hemiblock (bifascicular block)
* Uncontrolled hypertension
* Concomitant use of drugs with a risk of prolonging the QT interval or inducing torsades de pointes
* Concomitant use of CYP3A4 inhibitors
* Patients with unresolved diarrhea > CTCAE grade 1
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
* Other concurrent severe and/or uncontrolled medical conditions
* Patients who have received chemotherapy, any investigational drug or undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Concomitant use of any other anti-cancer therapy or radiation therapy
* Patients being treated with Coumadin (unless patients who require anticoagulation can be switched to a low-molecular weight or standard heparin)
* Female patients who are pregnant or breast feeding or patients of reproductive potential not willing to use a double method of contraception including a barrier method (i.e. condom) during the study and 3 months after the end of treatment (Women of childbearing potential [WOCBP] must have a negative serum pregnancy test within 7 days of the first administration of oral LBH589)
* Male patients whose sexual partners are WOCBP not willing to use a double method of contraception including condom during the study and 3 months after the end of treatment
* Patients with a history of another primary malignancy within 5 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-05; Primary Completion 2013-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of histone deacetylase inhibitor LBH589 in combination with imatinib mesylate | 1 month
Safety and tolerability of histone deacetylase inhibitor LBH589 in combination with imatinib mesylate | 4 months

SECONDARY OUTCOMES:
Effect of treatment with histone deacetylase inhibitor LBH589 in combination with imatinib mesylate on cytogenetic response status and BCR-Abl levels | 4 months
Effect of treatment with histone deacetylase inhibitor LBH589 in combination with imatinib mesylate on residual BCR-Abl positive primitive progenitors | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Bhatia, MD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - South Pasadena Cancer Center, South Pasadena, California
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington